CLINICAL TRIAL: NCT05892627
Title: PoZibio a Post-biotic Supplement on Cognitive Function and Brain Activity in Middle Age and Older Healthy Adults
Brief Title: A Supplement on Cognitive Function and Brain Activity in Middle Age and Older Healthy Adults
Acronym: PZAC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aberystwyth University (Other)
Collaborators: AGROCEUTICAL PRODUCTS LTD (Unknown); Neurodyn Life Sciences Inc. (Unknown); Postbiotics Inc (Unknown); Welsh Government (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 23766
Record Dates: First submitted 2023-04-28; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-04

CONDITIONS: Cognitive Decline
Keywords: Electroencephalography; Post-biotic; Lactobacillus paracasei; Cognitive health; Mental function; Metabolomics
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: A cohort who will be randomised into PoZibio™ (2 x capsules daily) or placebo (2 x capsules daily) supplementation for 6 weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PoZibio (Experimental): PoZibio, twice daily (50 x 10^9 CFUs/ CAPSULE) for 6 weeks
  Interventions: Dietary Supplement: PoZibio
- Placebo (Placebo Comparator): Placebo, twice daily for 6 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: PoZibio — PoZibio (50 x 10^9 CFUs/ CAPSULE)
  Arms: PoZibio
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
PoZibio™ capsules contains Lactobacillus paracasei which has been heat-killed (post-biotic).

The researchers will recruit a cohort of middle aged and older adults (>50 years) who will be randomised into PoZibio™ (2 x capsules daily) or placebo (2 x capsules daily) supplementation for 6 weeks. Subjects will be asked to take both capsules in the morning with their breakfast. The placebo will be matched to the active product by taste and texture.

Electroencephalography (EEG) shall be combined with 3 psychological tasks, to measure a variety of cognitive domains including attention, processing speed, accuracy, and response inhibition. These psychological tasks shall include the Stroop task, the Go/No-go task, and the Flanker task. Before taking part in the psychological tasks, participants shall be required to have their EEG resting state recorded, requiring them to participate in an Eyes Open/Closed Task.

The Mini Mental State Exam (MMSE) questionnaire shall be used as a digital screening tool to assess global cognitive function in participants both prior to and following the 6-week PoZibio trial. The geriatric depression scale (GDS) shall also be used as a digital screening tool to assess for depressive symptomatology in older adults. The EQ-5D questionnaire shall be used to obtain an overall profile of the health state and quality of life of participants before and after the trial.

The researchers will collect venous blood samples for the investigation into the chemical composition using metabolomics, the quantification of short chain fatty acids as well as clinical biochemistry, before and after the trial.

Aim:

A randomised, placebo controlled parallel human clinical trial of heat-treated Lactobacillus paracasei (post-biotics) in healthy middle aged and older subjects is proposed, to assess the potential for clinically relevant benefits in terms of cognitive function.

DETAILED DESCRIPTION:
Nowadays, the oral use of probiotics is widespread, in foods (i.e., yogurt), drinks (i.e., kombucha) and supplements. Heat-treated probiotics (essentially pasteurised or killed), cell-free supernatants, and purified key components can confer beneficial effects, mainly immune effects, protection against bacterial infections, and maintenance of gut health, which can positively impact on mental health and cognitive ability. Postbiotics, as they are called, have an advantage for food industry applications as they can easily be supplemented in several food lines/products and are shelf stable. PoZibio™ capsules contains the probiotics Lactobacillus paracasei which is a species of lactic acid bacteria often used in the fermentation of dairy products. It's found in the human intestinal tract and mouth, but also in foods such as yogurt and naturally fermented vegetables and milk. This has been heat-killed in PoZibio™(post biotic).

The researchers are aiming to recruit a cohort of middle aged and older adults (>50 years) who will be randomised into PoZibio™ (2 x capsules daily) or placebo (2 x capsules daily) supplementation for 6 weeks. Subjects will be asked to take both capsules in the morning with their breakfast. The placebo will be matched to the active product by taste and texture.

Electroencephalography (EEG) shall be combined with 3 psychological tasks in a computer program called E-Prime, to measure a variety of cognitive domains including attention, processing speed, accuracy, and response inhibition. These psychological tasks shall include the Stroop task, the Go/No-go task, and the Flanker task. Before taking part in the psychological tasks, participants shall be required to have their EEG resting state recorded, requiring them to participate in an Eyes Open/Closed Task.

The Mini Mental State Exam (MMSE) questionnaire shall be used as a digital screening tool to assess global cognitive function in participants both prior to and following the 6-week PoZibio™ trial. The geriatric depression scale (GDS) shall also be used as a digital screening tool to assess for depressive symptomatology in older adults. The EQ-5D questionnaire shall be used to obtain an overall profile of the health state and quality of life of participants, before and after the trial.

The researchers will collect venous blood samples for the investigation into the chemical composition using metabolomics, the quantification of short chain fatty acids as well as clinical biochemistry, before and after the trial.

Aim:

A randomised, placebo controlled parallel human clinical trial of heat-treated Lactobacillus paracasei (post-biotics) in healthy middle aged and older subjects is proposed, to assess the potential for clinically relevant benefits in terms of cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 50 years of age
* Subjects with Mini-Mental State Exam (MMSE) of 25-30 inclusive (global cognitive function)
* Subjects who are able to undergo EEG and to commit to visits to WARU/P5.
* Subjects who are able to provide venous blood samples.
* Subjects able to provide written informed consent PRIOR to performing any study procedures.

Exclusion Criteria:

* Subjects with diagnosis of Alzheimer's disease or other dementia
* Subjects taking medication for the treatment of dementia (such as acetylcholinesterase inhibitors (Aricept, Excelon), memantine (Namenda) or other medications with similar mechanisms of action) or medical foods (such as Cerefolin, Souvenaid, Axona) for the treatment of dementia.
* Subjects who are already regularly taking probiotics, post-biotics, nutraceutical and/or vitamin supplements related to PoZibio ™ within 30 days of screening.
* Subjects with Geriatric Depression Scale > 6
* Subjects with a Mini Mental State Exam score below 25
* Subjects who are pregnant or lactating
* Subjects with medical condition or disease that is life threatening
* Subjects who smoke cigarettes or use other products containing nicotine.
* Subjects diagnosed with diabetes.
* Subjects taking warfarin.
* Subjects who identify as being vegetarian or vegan
* Subjects who have a diagnosed or suspected mental health condition, or who have any concerns surrounding their mental health
* Subjects who have immediate family members with diagnosed mental health condition or suspected mental health concerns

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Control (Selective attention, processing speed, mental flexibility) | Improved score (faster response time and improved accuracy) from baseline score at 6 weeks after pozibio
  Cognitive Control (Selective attention, processing speed, mental flexibility) measured using the Stroop task in E-Prime
Cognitive Control (Selective attention, processing speed, mental flexibility) | Improved score (faster response time and improved accuracy) at 6 weeks after pozibio when compared with placebo after 6 weeks
  Cognitive Control (Selective attention, processing speed, mental flexibility) measured using the Stroop task in E-Prime
Response inhibition (core construct in cognitive control and self-regulation) | Improved (fewer commission errors) score from baseline score at 6 weeks after pozibio
  Measured using the Go/No-go task in E-Prime
Response inhibition (core construct in cognitive control and self-regulation) | Improved (fewer commission errors ) score at 6 weeks after pozibio when compared with placebo after 6 weeks
  Response inhibition (core construct in cognitive control and self-regulation) measured using the Go/No-go task in E-Prime
Selective attention and response inhibition (core constructs in cognitive control and self-regulation) | Improved score (faster response time and improved accuracy) from baseline score at 6 weeks after pozibio
  Selective attention and response inhibition (core constructs in cognitive control and self-regulation) measured using the Flanker task in E-Prime
Selective attention and response inhibition (core constructs in cognitive control and self-regulation) | Improved score (faster response time and improved accuracy) at 6 weeks after pozibio when compared with placebo after 6 weeks
  Selective attention and response inhibition (core constructs in cognitive control and self-regulation) measured using the Flanker task in E-Prime
Electroencephalogram (EEG) during the Stroop task | After 6 weeks of pozibio, no delay of the P3 component and more N2 components when compared with baseline
  Assessing event related potentials (ERP's) in the P3 component and the N2 component across the frontal and parietal regions
Electroencephalogram (EEG) during the Stroop task | After 6 weeks of pozibio, no delay of the P3 component and more N2 components when compared with 6 weeks of placebo
  Assessing event related potentials (ERP's) in the P3 component and the N2 component across the frontal and parietal regions
Electroencephalogram (EEG) during the Flanker task | After 6 weeks of pozibio, no delay of the P3 component and more N2 components when compared with baseline
  Assessing event related potentials (ERP's) in the P3 component and the N2 component across the frontal and parietal regions
Electroencephalogram (EEG) during the Flanker task | After 6 weeks of pozibio, no delay of the P3 component and more N2 components when compared with 6 weeks of placebo
  Assessing event related potentials (ERP's) in the P3 component and the N2 component across the frontal and parietal regions
Electroencephalogram (EEG) during the go/no-go task | After 6 weeks of pozibio, no delay of the P3 component and more N2 components when compared with baseline
  Assessing event related potentials (ERP's) in the P3 component and the N2 component across the frontal and parietal regions
Electroencephalogram (EEG) during the go/no-go task | After 6 weeks of pozibio, no delay of the P3 component and more N2 components when compared with 6 weeks of placebo
  Assessing event related potentials (ERP's) in the P3 component and the N2 component across the frontal and parietal regions
Electroencephalogram (EEG) during the stroop task | After 6 weeks of pozibio, increased alpha and delta activity when compared with baseline
  Assessing alpha and delta activity
Electroencephalogram (EEG) during the Flanker task | After 6 weeks of pozibio, increased alpha and delta activity when compared with baseline
  Assessing alpha and delta activity
Electroencephalogram (EEG) during the go/no-go task | After 6 weeks of pozibio, increased alpha and delta activity when compared with baseline
  Assessing alpha and delta activity
Electroencephalogram (EEG) during the stroop task | After 6 weeks of pozibio, increased alpha and delta activity when compared with 6 weeks of placebo
  Assessing alpha and delta activity
Electroencephalogram (EEG) during the Flanker task | After 6 weeks of pozibio, increased alpha and delta activity when compared with 6 weeks of placebo
  Assessing alpha and delta activity
Electroencephalogram (EEG) during the go/no-go task | After 6 weeks of pozibio, increased alpha and delta activity when compared with 6 weeks of placebo
  Assessing alpha and delta activity
EuroQol 5 Dimension 5L (combined score) | Reduced score from baseline EuroQol 5 Dimension 5 score at 6 weeks after pozibio
  EuroQol 5 Dimension 5 5L questionnaire: Generic quality of life. Mobility- Level 1-5 Self-Care- Level 1-5, Usual Activities- Level 1-5, Pain/Discomfort- Level 1-5, Anxiety/Depression- Level 1-5. The digits for the five dimensions will be combined into a 5-digit number that describes the patient's health state.
EuroQol 5 Dimension 5L (combined score) | Reduced EuroQol 5 Dimension 5 score at 6 weeks after pozibio when compared with placebo after 6 weeks
  EuroQol 5 Dimension 5 5L questionnaire: Generic quality of life. Mobility- Level 1-5 Self-Care- Level 1-5, Usual Activities- Level 1-5, Pain/Discomfort- Level 1-5, Anxiety/Depression- Level 1-5. The digits for the five dimensions will be combined into a 5-digit number that describes the patient's health state.

SECONDARY OUTCOMES:
Changes in short chain fatty acids concentrations in plasma | Increased concentration of total short chain fatty acids after the pozibio at 6 weeks compared with the baseline
  Changes in short chain fatty acids concentrations in plasma measured using Gas Chromatography-Flame Ionization Detection
Changes in short chain fatty acids concentrations in plasma | Increased concentration of total short chain fatty acids after the pozibio at 6 weeks compared with that after placebo at 6 weeks
  Changes in short chain fatty acids concentrations in plasma measured using Gas Chromatography-Flame Ionization Detection

CONTACTS AND LOCATIONS:
Overall Officials: Amanda J Lloyd, PhD, BSc, Principal Investigator — Aberystwyth University
Locations (1):
- Well-being and Health Assessment Research Unit (WARU), Aberystwyth, Ceredigion, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available to other researchers

DOCUMENTS (1):
  • Study Protocol (2023-05-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT05892627/Prot_000.pdf